CLINICAL TRIAL: NCT06140225
Title: Promotion of Daily Recommended Physical Activity for Adolescents' Health Through Mobile Apps, Wearables, and a Gamified TAC
Brief Title: Adolescents' Health Through Mobile Apps, Wearables, and a Gamified TAC ( ActivA-App )
Acronym: ActivA-App
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Raquel Vaquero-Cristóbal, Principal investigator, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Project ActivA-App; PID2022-140245OA-I00 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación)
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Adolescent Behavior; Physical Activity; New Technologies
Keywords: Adolescents; Physical activity; New Technologies; Psychology
MeSH Terms: conditions — Adolescent Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- "PACER" Application (Experimental): It is an application that allows the recording of the sports activities performed. It includes alerts and reminders that allow the participant to plan his/her sports practice in advance, as well as a weekly record of the activities and kilometers run, and a comparative analysis with the previous week.
  Interventions: Behavioral: "PACER" Application
- "MapMyWalk" Application (Experimental): It is an application that promotes the practice of physical activity by recording the sports activities that the subject performs, as well as the dissemination of the same in social networks and participation in challenges available to users around the world. In addition, this application includes reminders of physical activity and personal achievements to encourage the practice of sports.
  Interventions: Behavioral: "MapMyWalk" Application
- "Strava" Application (Experimental): It is an application that promotes sports practice, nutritional habits and the necessary rest. Nutrition and sleep will be introduced as variables that favor a healthy lifestyle
  Interventions: Behavioral: "Strava" Application
- "POKEMON GO" APPLICATION (Experimental): It is a mobile game that favors the increase of physical activity because it is necessary to walk to achieve the proposed objectives.
  Interventions: Behavioral: "POKEMON GO" APPLICATION
- "JEFIT" APPLICATION (Experimental): It is an app whose goal is to be a support in training of strength-resistance training. Setting a specific goal, with a full databaseover of exercises to perform.
  Interventions: Behavioral: "JEFIT" APPLICATION
- "FITBIT-FLEX" APPLICATION (Experimental): It is a physical activity wereable. It acts as a witness to physical activity and transmits the data to the computer or smartphone.
  Interventions: Behavioral: "FITBIT-FLEX" APPLICATION
- "MEIZU BONG 2S" APPLICATION (Experimental): It is a physical activity wereable. It acts as a witness to physical activity and transmits the data to the computer or smartphone.
  Interventions: Behavioral: "MEIZU BONG 2S" APPLICATION
- Control Group (No Intervention): They will not use any type of sports technology application. They will continue to perform their daily activities without intervention.

INTERVENTIONS:
Behavioral: "PACER" Application — It is an application that allows the recording of the sports activities performed. It includes alerts and reminders that allow you to plan your sports practice in advance, as well as a weekly record of the activities and kilometers run, and a comparative analysis with the previous week.
  Arms: "PACER" Application
Behavioral: "MapMyWalk" Application — It is an application that promotes the practice of physical activity by recording the sports activities that the subject performs, as well as the dissemination of the same in social networks and participation in challenges available to users around the world. In addition, this application includes reminders of physical activity and personal achievements to encourage the practice of sports.
  Arms: "MapMyWalk" Application
Behavioral: "Strava" Application — It is an application that promotes sports practice, nutritional habits and the necessary rest. Nutrition and sleep will be introduced as variables that favor a healthy lifestyle.
  Arms: "Strava" Application
Behavioral: "POKEMON GO" APPLICATION — It is a mobile game that favors the increase of physical activity because it is necessary to walk to achieve the proposed objectives.
  Arms: "POKEMON GO" APPLICATION
Behavioral: "JEFIT" APPLICATION — It is an app whose goal is to be a support in training of strength-resistance training. Setting a specific goal, with a full databaseover of exercises to perform.
  Arms: "JEFIT" APPLICATION
Behavioral: "FITBIT-FLEX" APPLICATION — It is a physical activity wereable. It acts as a witness to physical activity and transmits the data to the computer or smartphone.
  Arms: "FITBIT-FLEX" APPLICATION
Behavioral: "MEIZU BONG 2S" APPLICATION — It is a physical activity wereable. It acts as a witness to physical activity and transmits the data to the computer or smartphone.
  Arms: "MEIZU BONG 2S" APPLICATION

SUMMARY:
A primary factor in preventing diseases in adulthood, as well as overweight and obesity, is the promotion of physical activity from childhood and adolescence. Although the recommendations for practicing physical activity at this stage are broad, low rates of practice that do not comply with the recommendations are reported. There is a high percentage of use of new technologies, particularly mobile applications, they have been used with some success to improve the health of similar populations, although its use for this purpose has certain limitations. Therefore, this project will investigate whether the use of various mobile and wearable applications can be an effective way to periodically increase physical activity levels and establish new healthy habits that improve the present and future health of adolescents. Several secondary education centers in the Region of Murcia will participate in this project. The objective is to obtain relevant results that can serve as a starting point for other interventions at a national or international level.

DETAILED DESCRIPTION:
The promotion of physical activity among young people has become a crucial factor in preventing adult-onset diseases, particularly overweight and obesity, and in improving health and well-being during this stage. The World Health Organization (WHO) recommends 60 minutes of moderate aerobic activity per day (or the equivalent in vigorous activity) and at least three days a week of strength-resistance exercises for children and adolescents. However, surveys on the physical activity habits of Spanish adolescents indicate that more than 50% do not meet these recommendations. Excessive use of new technologies has been identified as a predisposing factor for decreased physical activity, a habit that is increasingly common among adolescents. This, combined with the sedentary conditions brought about by the COVID-19 pandemic, has led to a significant increase in sedentary behavior among the young population. Nevertheless, new technologies, particularly mobile applications, have been used with some success to improve the health of similar populations, although their use for this purpose has certain limitations. Therefore, this project aims to address the decline in physical activity among the adolescent population and provide resources that will endure over time to promote physical activity among adolescents within the educational sphere. It's worth noting that during the period of Compulsory Secondary Education (ESO), there are only two hours of Physical Education (PE) per week, making it impossible to meet the recommended levels of practice solely through school-based physical activity. Thus, it is necessary to create resources that encourage physical activity in leisure time, involving both students and teachers, and that can also be utilized by future generations. This project builds upon prior research in promoting physical activity through Information and Communication Technologies (ICTs), but adapts it to a more sedentary social context, vastly different from before, requiring new strategies to increase physical activity in adolescents and thereby promote the preservation of physical and mental health following the inactivity imposed by the COVID-19 lockdown. Therefore, this project will investigate whether the use of various mobile applications and wearables can be an effective way to regularly increase physical activity levels and establish new healthy habits that improve both present and future health for adolescents. Additionally, it aims to provide teachers and students with an application that effectively encourages physical activity within the educational context, guided by professionals in Physical Activity and Sports Sciences, yet remains engaging and motivating for continued use. This will allow for a combination of physical activity and education within the context of Technology-Enhanced Learning and Communication (TAC). This project will involve several secondary education centers in the Region of Murcia, as it is one of the autonomous communities with higher levels of inactivity, overweight, and obesity in early ages. The goal is to obtain relevant results that can serve as a starting point for other interventions at a national or international level.

ELIGIBILITY:
Inclusion Criteria:

* Be a student of compulsory secondary education
* Not present any disease or surgical operation that would prevent the performance of the physical tests or the follow-up of the established intervention.
* Complete the questionnaires provided and carry out the established tests in their entirety
* Have access to any mobile device that allows access to the technological sports applications used in the intervention.

Exclusion Criteria:

* Failure to complete the questionnaires provided and/or to take the prescribed tests in their entirety
* Failure to complete scheduled intervention activities.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Level (International Physical Activity Questionnaire for Adolescents) | Pre-test, week 10, week 20 and week 24
  The PAQ-A (Martínez-Gómez et al., 2009) will be used to establish the level of sports practice of the adolescents. This questionnaire includes eleven questions related to the practice of physical activity in school, after school, household chores and travel. The questionnaire makes it possible to classify adolescents as inactive or active (light, moderate or vigorous intensity). The questionnaire reports the time in hours and minutes that the participant performs physical activity. The longer the time, the better the result.
Physical activity level (accelerometry) | Pre-test, week 10, week 20 and week 24
  In a subset of secondary school students (n=30), physical activity will be analyzed using accelerometry with the Actigraph GT3X+Tri-Axis Accelerometer Monitor (Actigraph, Pensacola, Florida). To do this, participants will be asked to wear the accelerometer on their non-dominant hand continuously for seven consecutive days and nights. They will be instructed not to move the accelerometer during the measurement period (Hjorth et al., 2012).
Use of internet (CERI Questionnaire) | Pre-test, week 10, week 20 and week 24
  To measure the frequency of Internet use through new communication technologies, the CERI questionnaire (Fargues et al. 2009) will be used, which includes 10 questions rated on a scale of 1 to 4, with 1 being "almost never" and 4 "almost always". The questionnaire reports a number from 10 to 40, with the higher value being more use.
Use of mobile phone (CERM Questionnaire) | Pre-test, week 10, week 20 and week 24.
  To measure the frequency of cell phone use, regardless of whether it is for social networks, video games, etc., the CERM questionnaire (Fargues et al. 2009) will be used, which includes 10 questions rated on a scale of 1 to 4, with 1 being "almost never" and 4 being "almost always". The questionnaire reports a number from 10 to 40, with the higher value being a more use.
Satisfaction with life (Life Satisfaction Scale) | Pre-test, week 10, week 20 and week 24
  Life satisfaction is defined as a person's overall evaluation of his or her life. The person examines the tangible aspects of his or her life and compares them with a standard or criterion chosen by him or her, arriving at a judgment about satisfaction with his or her life (Pavot et al., 1991). Thus, judgments about satisfaction depend on the comparisons the subject makes between the circumstances of his or her life and a standard that he or she considers appropriate. The life satisfaction scale (Diener et al., 1985) provides information on feelings of happiness, feelings of loneliness and satisfaction in school among adolescents, obtaining an overall assessment of life satisfaction. The scale is composed of five questions that are answered on a scale of 1 to 5, with 1 being "strongly disagree" and 5 "strongly agree". The minimum score will be 5 and the maximum 25 points. A higher score indicates greater satisfaction with life.
Physical condition (Maximal oxygen consumption) | Pre-test, week 10, week 20 and week 24
  The 20-m shuttle run test evaluates maximal aerobic capacity by means of an incremental 20-meter out-and-back test. The initial speed of the test is 8.5 km/h and is increased every minute by an audible signal. The test ends when the subject stops or fails to reach the reference line two consecutive times. The speed recorded is the speed reached in the last stage that the subject is able to complete. Through the equations of Leger, Mercier, Gadoury and Lambert (1988) the reference value of the subject's VO2 max. is obtained.
Physical condition (Handgrip Strength) | Pre-test, week 10, week 20 and week 24
  The test will provide information about the isometric force (kg) that the participant is able to develop with the forearm musculature. For this purpose, a digital dynamometer with manual grip (5030J1, Jamar ®, Sammons Preston, United Kingdom) will be used. Prior to the execution, the instrument will be adjusted according to the age of the player and the length of his/her hand. Two measurements will be taken with each arm, with a one minute rest between them. The participant must hold the dynamometer with the executing hand and the arm extended along the torso, without contacting it, and produce the maximum force possible (Rojas, Vázquez, Sánchez, Banik, & Argáez, 2012; Valdes & Yanci, 2016). Manual grip strength determined by dynamometer is significantly associated with proper cardiovascular health in adolescents, so its analysis is of interest as part of an assessment of global physical fitness (García-Hermoso et al., 2019).
Physical condition (Lower extremity muscle strength) | Pre-test, week 10, week 20 and week 24
  The countermovement jump test (CMJ) will be used to measure this variable. This test provides information on the explosive strength of the lower body. The CMJ is a vertical jump that begins with the subject in a standing position, followed by knee flexion to a position of approximately 90 degrees, and a rapid extension of the knees to perform a jump in which the maximum height is reached. It should be noted that there is no stop in the knee flexion position since the intention is to take advantage of the explosive elastic reflex energy of the movement. The subjects will perform two repetitions of the jump 2 minutes apart. A MuscleLab force platform (Ergotest Innovation S.A., Norway) will be used to record the data, which will measure the time of flight from the time the subject takes off from the platform to the time the subject re-enters contact with the platform.
Physical condition (Hamstrings Flexibility) | Pre-test, week 10, week 20 and week 24
  The sit-and-reach test will be used. A 30-centimeter measuring box (Finder Flex-Tester, Novel Products, USA) with a millimeter ruler is required. In the initial position, the subject should be in a seated position, with knees fully extended feet hip-width apart and soles of the feet perpendicular to the floor and in contact with the box. The subject will be asked to place one hand on top of the other, with the palms of the hands facing downward and the fingers stretched out. The subject will perform a neck flexion to bring the chin to the chest and a trunk flexion with the knees fully stretched and without ballistic movements, trying to reach the greatest possible distance and maintaining the posture for 3 seconds. The distance will be measured in centimeters and the value 0 will correspond to the tangent of the soles of the feet, the values being positive when this distance is exceeded, and negative when it is not reached.
Physical condition (horizontal jump) | Pre-test, week 10, week 20 and week 24.]
  Upper lower body strength is measured form a standing position with feet approximately shoulder´s width apart. Participant jump as far forward as possible. The test is performance twice. The longest distance achieved was recorded in centimeters20.
Anthropometric Variables (Height) | Pre-test, week 10, week 20 and week 24
  To measure height, a SECA measuring rod should be used. Adolescents should stand barefoot with their backs against the measuring rod, heels of their feet together and their gaze straight ahead. Measurements will be obtained in centimeters and will be repeated 2 times for each subject. A third measurement will only be taken if the difference between the first and second measurement is greater than 1%.
Anthropometric Variables (Weight) | Pre-test, week 10, week 20 and week 24.]
  A Tanita BC 418-MA Segmental scale (Tanita, Tokyo) will be used to measure body weight. The subject will step on the scale with both feet inside the scale and looking straight ahead, without leaning the body. Values will be obtained in kilograms and two measurements will be carried out on each subject. If the difference between both measurements is greater than 1%, a third measurement will be taken
Anthropometric Variables (Fat mass) | Pre-test, week 10, week 20 and week 24.
  To obtain the fat mass, it will be necessary to previously measure the triceps, thigh and leg folds, and the waist, hip, relaxed arm, thigh and leg perimeters. For these previous measurements, two measurements will be taken in each subject, and a third measurement will be necessary if the difference between the first two is greater than 5%. Once the values of the previous measurements have been obtained, the fat mass can be calculated using the formula of Slaughter et al. (1988)
Anthropometric Variables (Fat-free mass) | Pre-test, week 10, week 20 and week 24.
  To obtain the fat-free mass, it will be necessary to previously measure the triceps, thigh and leg folds, and the perimeters of the waist, hip, relaxed arm, thigh and leg. For these previous measurements, two measurements will be taken in each subject, and a third measurement will be necessary if the difference between the first two is greater than 5%. Once the values of the previous measurements have been obtained, the-fat free mass can be calculated using the formula of Poortmans et al. (2005)
Physical condition (upper limb strength) | Pre-test, week 10, week 20 and week 24
  To assess upper limb strength will be used Push-up test. The subject will perform as many repetitions as possible in one minute, or until reaching exhaustion (Castro-Piñero et al., 2010).
Physical condition (Curl-up) | Pre-test, week 10, week 20 and week 24
  To assess abdominal muscle endurance will be use Curl-up. The highest number of repetitions the subject completes in one minute will be recorded (García-Pastor et al., 2016).
Physical condition (Maximum speed) | Pre-test, week 10, week 20 and week 24.
  To assess maximum speed will be used 20-m sprint. A maximum speed sprint over 20 meters will be performed, following the protocol of previous research (García-Manso et al., 1996). Photocells placed at hip height will be used for timing quantification (Altmann et al., 2017).
Anthropometric Variables (BMI) | Pre-test, week 10, week 20 and week 24.
  Previously obtained height and weight measurements will be used to establish the BMI. The formula used will be weight/height^2, and the result will be obtained in kg/m^2. This index is commonly used and is related to metabolic and cardiovascular diseases in adolescents and adults.
Satisfaction and frustration of basic psychological needs | Pre-test, week 10, week 20 and week 24.
  This questionnaire is made up of 24 items grouped into six factors and analyze different basic psychological needs, as described in the Self-Determination Theory (SDT), developed by Deci and Ryan. Autonomy is evaluated by four items, relatedness is evaluated by four items, and competence by four items. The frustration of each of the basic psychological needs, in turn, is evaluated by four elements each. The 14 items will be evaluated through a five-point Likert-type scale, ranging from 1 (completely false) to 5 (completely true). All factors values range 4 and 20 points. Higher scores report a better score in the factor.
Motivation in Physical Education Classes | Pre-test, week 10, week 20 and week 24.
  To assess motivation towards physical education classes, the Perceived Locus of Causality Scale (PLOC) has been used. This scale is made up of 20 items on a 7-point Liker scale from completely agree to completely disagree. These items evaluate 5 factors: intrinsic motivation, identified regulation, introjected regulation, external regulation and amotivation. All factors values range 1 and 7 points. Higher scores report a better score in the factor.
Fat percentage | Pre-test, week 10, week 20 and week 24.
  It will assessed by bioimpedance in percentage, following the recommendations of Brantlov et al. (2017) for proper execution.
Hydration percentage | Pre-test, week 10, week 20 and week 24.
  It will assessed by bioimpedance in percentage, following the recommendations of Brantlov et al. (2017) for proper execution.
Muscle mass | Pre-test, week 10, week 20 and week 24.
  It will assessed by bioimpedance in kilogramers, following the recommendations of Brantlov et al. (2017) for proper execution.
Bone weight | Pre-test, week 10, week 20 and week 24.
  It will assessed by bioimpedance, in kilogramers, following the recommendations of Brantlov et al. (2017) for proper execution.
Visceral fat | Pre-test, week 10, week 20 and week 24.
  It will assessed by bioimpedance in kilogramers, following the recommendations of Brantlov et al. (2017) for proper execution.

SECONDARY OUTCOMES:
Healthy lifestyle habits (Survey on Healthy Habits in Adolescents) | Pre-test, week 10, week 20 and week 24
  The "Survey on Healthy Habits in Adolescents" (ENHASA) will be used. This questionnaire consists of 26 items that are completed using a Likert scale of 0-10 points, addressing four dimensions related to the main risk factors: nutrition, physical activity, new technologies, and environment. The final score allows for the following classification: very poor habits, poor, acceptable, good, and very good (Carpena-Lucas et al., 2022; Jiménez-Candel et al., 2021).
Evaluation of ICTs (User version of the Mobile Application Rating Scale) | week 10
  The User version of the Mobile Application Rating Scale (uMARS) is a scale consisting of 26 items completed using a Likert scale ranging from 1 to 5 points. This scale allows for the assessment of 6 dimensions, which include engagement, functionality, aesthetics, information, subjective quality, and perceived impact of the mobile application (Martin-Payo et al., 2021). All factors values range 1 and 5 points. Higher scores report a better score in the factor
Biological maturation | Pre-test, week 10, week 20 and week 24.
  Biological maturation will also be assessed since it can be crucial during this stage of development. To do this, the sexspecific formula from Mirwald et al. (2002) will be used to estimate the maturation offset of the adolescents. Based on the maturation offset, the biological maturation of each subject will be calculated (Albaladejo-Saura et al., 2022).
Academic performance | Week 10, week 20 and week 24.]
  The educational institution will be asked for the academic record of the academic year in which the measurements are conducted for the participating students in order to establish the relationship between the level of physical activity and academic performance. Academic performance will be obtained with the average grade of all the subjects taken by the participant in the course in which the program is developed. This average grade will be provided by the school.
Mediterranean Diet Quality (KIDMED Questionnaire) | Pre-test, week 10, week 20 and week 24
  The KIDMED questionnaire (Serra-Majem et al., 2004) will be used to establish the level of adherence of adolescents to the Mediterranean diet. It consists of 16 questions that are scored with a value of -1 if they denote a negative connotation with respect to the Mediterranean diet, or with a +1 if they are positive in relation to the diet. The index ranges from 0 to 12 points and the results are classified as: optimal Mediterranean diet (>8 points), requires improvement to adjust intake to Mediterranean patterns (4-7 points), and very low diet quality (≤ 3 points). The questions included in the questionnaire are related to the main foods included in this type of diet (fruit, vegetables, bread, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Vaquero-Cristobal, PhD, Principal Investigator — Universidad de Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mateo-Orcajada A, Abenza-Cano L, Vaquero-Cristobal R. Protocol for a randomized controlled trial of a mobile app and wearable-based intervention promoted through physical education to enhance physical and psychological health in adolescents during out-of-school hours. BMC Public Health. 2025 Dec 26;26(1):359. doi: 10.1186/s12889-025-25919-8. PMID 41454278